CLINICAL TRIAL: NCT02812823
Title: Comparison of High-resolution Anorectal Manometry and 3D High-definition Anorectal Manometry in Diagnosis of Functional Disorders in Children
Brief Title: Comparison of Anorectal Manometry and 3D Manometry in Diagnosis of Functional Disorders in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Marcin Banasiuk, PhD, Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Banasiuk 2016A
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Constipation; Children; Fecal Incontinence
Keywords: manometry; children; constipation; functional disorders
MeSH Terms: conditions — Constipation; Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High resolution anorectal manometry (Other): All subjects will be investigated by high-resolution anorectal manometry. At the beginning the anorectal cather will be used to record conventional parameters and after that 3D high-definition anorectal manometric catheter will be inserted in order to measure conventional parameters and 3D picture of anorectum.
  Interventions: Device: High-resolution anorectal manometry

INTERVENTIONS:
Device: High-resolution anorectal manometry — Recording of conventional manometric parameters after insertion of the catheters.

SUMMARY:
Pressures measured by manometric solid-state catheters may differ according to the type of the catheter and specific anatomy and physiology of anorectum.

The aim of the study is to establish the difference in recordings between 2 types of anorectal catheters used in pediatric patients and to validate the most appropriate way to diagnose of functional disorders.

DETAILED DESCRIPTION:
Patients enrolled in study will be investigated by both types of anorectal catheters, first by anorectal high resolution flexible, thinner, solid-state catheter and after that with rigid, thicker, solid-state catheter. Both procedures will be undertaken during one session. There will be used standard protocol of the procedure that measures conventional manometric parameters (resting pressure, squeeze pressure, bear down manoeuver, thresholds of sensation and recto anal inhibitory reflex threshold.

ELIGIBILITY:
Inclusion Criteria:

* Functional Constipation
* Fecal Incontinence
* Parental Agreement

Exclusion Criteria:

* After surgery on lower gastrointestinal tract
* Diagnosis of inflammatory bowel disorders
* Diagnosis of other disorders present in anorectal area, that may influence anorectal pressures
* Lack of parental agreement

Ages: 4 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Difference in Resting pressure of the anorectal area | 20 seconds
  Resting pressure will be measured after insertion catheter into anorectum. The software automatically record pressure while patient is lying on the bed.
  The parameter is recorded with 2 different types of anorectal catheters and the difference is evaluated.

SECONDARY OUTCOMES:
Maximum squeeze pressure | 1 min
  Pressure is recorded after the patient is asked to squeeze anorectum for 20 s (repeated 3 times).
Bear down manoeuver | 1 min
  Pressures are recorded after the patient is asked to bear down for 20 s (repeated 2 times)
Thresholds of sensation | 1 min
  The balloon at the top of the catheter is being filled with air until a patient is able to report sensation, urge and discomfort.
Recto anal inhibitory reflex | 5 min
  The balloon at the top of the catheter is being filled with air until the relaxation of anal sphincter is observed.

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Banasiuk, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Pediatric Gastroenterology and Nutrition, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banasiuk M, Dobrowolska ME, Skowronska B, Konys J, Banaszkiewicz A. Comparison of Anorectal Function as Measured with High-Resolution and High-Definition Anorectal Manometry. Dig Dis. 2022;40(4):448-457. doi: 10.1159/000518357. Epub 2021 Aug 10. PMID 34515101